CLINICAL TRIAL: NCT02034851
Title: Phase 3- Dexamethasone Administration in 1st Episode of Febrile Urinary Tract Infection Episode as Renal Damage Prevention Strategy. DEXCAR
Brief Title: Dexamethasone Administration in 1st Episode of Febrile Urinary Tract Infection
Acronym: DEXCAR-0212
Status: Completed | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Hospital Universitari Sant Joan de Reus (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Pius Hospital de Valls (Unknown); Hospital Arnau de Vilanova (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Maternal-Infantil Vall d´Hebron Hospital (Other); Hospital General Universitario Santa Lucía (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor
Other Study IDs: IISPV_Pediatria_Dexcar; 2011-005805-66 (EudraCT Number)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2014-04

CONDITIONS: Acute Pyelonephritis
Keywords: Acute pyelonephritis; Renal scarring; Dexamethasone; Children; Corticoids; Complementary treatment; Prevention strategy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Dexamethasone: Intervention group
- Control: Placebo group (physiological saline)

SUMMARY:
Hypothesis: Administration of corticoids (dexamethasone) together with the conventional antibiotherapy in the acute phase of a febrile urinary tract infection could reduce the risk of renal scarring after 6 months of the primo-infection.

Primary objectives:To evaluate the reduction in incidence of renal scarring after 6 months of a acute pyelonephritis between the control group (conventional therapy plus placebo) and intervention group (conventional therapy plus dexamethasone.

Design: Multicentre randomized clinical trial,placebo controled, including children between 2 months and 14 years with a acute pyelonephritis proven by a acute phase DMSA (dimethylsuccinic acid ). A total of 180 children in to parallel groups (intervention and placebo) will be included.

DETAILED DESCRIPTION:
The urinary tract infection (UTI) is one of the most common bacterial infections in children. These infections can be grouped clinically as asymptomatic bacteriuria , cystitis (lower urinary tract infection ) and acute pyelonephritis (APN ) when the infection reaches the upper urinary tract. This classification is of great clinical relevance because while cystitis is usually a benign condition without further complications , the APN is associated with an increased risk of kidney damage, acquired through renal scarring . Renal scarring is a consequence of the inflammatory and immune response that is triggered to eradicate the bacteria involved in the UTI. Parenchymal infection can be solved , but there are a number of poorly understood factors that may perpetuate inflammation and this would promote the formation of scar nephritis. One of the most relevant factors involved in the renal scarring development are the production of inflammatory mediators (complement proteins, bactericidal peptides, cytokines such as IL6 and IL8, chemokines, and adhesion molecules defensins). Thus, it is obvious to think that the use of anti-inflammatory drugs may prevent the release of these mediators and the development of permanent kidney damage.

Intervention: the two parallel groups will receive the conventional therapy plus:

1. dexamethasone: 0'30 mg per kg every 12 hours during 3 days.
2. placebo (physiological saline)at the same dosing regimen.

Centralized lecture of the late DMSA after 6 months of the pyelonephritis episode will be performed. Renal scarring presence and grade will be reported.

ELIGIBILITY:
Inclusion Criteria:

Those children between 2 months and 14 years with a provable acute pyelonephritis that fulfill the hospitalization criteria defined in the Spanish Clinical practice guide. Briefly:

* age under 3 months.
* general affectation, toxic appearance.
* vomiting or oral intolerance.
* dehydration, bad peripheric perfusion.
* or other intermedia situations that include:

  1. high fever (>38.5 Celsius) in 3-6 month old children.
  2. unusual germ risk factors.
  3. family history of vesicoureteral reflux.
  4. recurrent febrile urinary infections. With absence of a previous renal scarring objectivated after a DMSA.
  5. high elevation of acute phase reactants.

Exclusion Criteria:

* those eligible patients that do not fulfill the hospitalization criteria.
* patients with a procalcitonin under 0.05 ng per ml.
* patients with previous uropathy or renal scarring
* patients allergic to dexamethasone.
* endocrinologic disease.
* history of cancer.
* serious illness.
* immunosuppressor treatment.
* previous treatment with corticoids (continuous oral or parenteral treatment) during the last 2 months.
* the patient included in the study that do not present pyelonephritis after the acute phase DMSA evaluation will be excluded.
* the patient included in the study that suffered a second pyelonephritis episode during the following 6 months (before the second DMSA evaluation) will be excluded for the primary output analyses.

Ages: 2 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Those children between 2 months and 14 years with a provable acute pyelonephritis that fulfill the hospitalization criteria defined in the Spanish Clinical practice guide.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
renal scarring | 6 month after the acute pyelonephritis episode

CONTACTS AND LOCATIONS:
Overall Officials: Escribano J Joaquin, PhD MD, Principal Investigator — IISPV- URV-Hospital Universitari Sant Joan de Reus- Research unit in pediatrics, nutrition and human development; Closa R Ricardo, MD PhD, Principal Investigator — IISPV-URV- Hospital Universitari Joan XXIII de Tarragona-Research unit in pediatrics, nutrition and human development; Ferré N Natalia, PhD, Principal Investigator — IISPV-URV-Research unit in pediatrics, nutrition and human development; Ibars Z Zaira, MD PhD, Study Director — HOSPITAL ARNAU DE VILANOVA DE LLEIDA; Maria Gloria MG Fraga, MD PhD, Study Director — HOSPITAL DE LA SANTA CREU I SANT PAU, DE BARCELONA; Madrid A Alvaro, MD PhD, Study Director — HOSPITAL MATERNOINFANTIL VALL D'HBRON, BARCELONA; Samper M Manuel, MD PhD, Study Director — Pius Hospital de Valls; Gonzalez JD Juan David, MD PhD, Study Director — HOSPITAL GENERAL UNIVERSITARIO SANTA LUCÍA DE CARTAGENA; Parada E Esther, MD PhD, Study Director — HOSPITAL JOAN XXII DE TARRAGONA
Locations (7):
- Spain (7):
  - Hospital General Universitario Santa Lucía de Cartagena, Cartagena, Murica
  - Iispv- Hospital Sant Joan de Reus, Reus, Tarragona
  - Pius Hospital de Valls, Valls, Tarragona
  - Hospital Maternoinfantil Vall D'Hebron, Barcelona
  - Hospital de La Santa Creu I Sant Pau de Barcelona, Barcelona
  - Hospital Arnau de Vilanova de Lleida, Lleida
  - Iispv-Hospital Joan Xxii de Tarragona, Tarragona

REFERENCES:
- [Derived] Rius-Gordillo N, Ferre N, Gonzalez JD, Ibars Z, Parada-Ricart E, Fraga MG, Chocron S, Samper M, Vicente C, Fuertes J, Escribano J; DEXCAR Study Group. Dexamethasone to prevent kidney scarring in acute pyelonephritis: a randomized clinical trial. Pediatr Nephrol. 2022 Sep;37(9):2109-2118. doi: 10.1007/s00467-021-05398-w. Epub 2022 Jan 18. PMID 35041042